CLINICAL TRIAL: NCT03922919
Title: Effect of Administration of 3rd Generation Cephalosporin (Ceftriaxone Versus Cefotaxime) on the Digestive Carrying of 3rd Generation Cephalosporin-resistant Enterobacteriaceae (EB C3G-R)
Brief Title: Effect of Administration of 3rd Generation Cephalosporin on the Digestive Carrying of 3rd Generation Cephalosporin-resistant Enterobacteriaceae (CEF-IMPACT)
Acronym: CEF-IMPACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: API/2016/74
Record Dates: First submitted 2019-02-21; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-02

CONDITIONS: Infectious Disease - Resistant Enterobacteriaceae (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Cefotaxime; Ceftriaxone

STUDY DESIGN:
Intervention Model Description: stepped-wedge design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefotaxime or ceftriaxone group (Active Comparator): free use of cefotaxime or ceftriaxone by the investigator
  Interventions: Procedure: Rectal swab; Drug: Cefotaxime/ceftriaxone
- Cefotaxim group (Experimental): Systematic use of cefotaxime
  Interventions: Drug: Cefotaxime Injection; Procedure: Rectal swab

INTERVENTIONS:
Drug: Cefotaxime Injection — Systematic use of cefotaxime.
  Arms: Cefotaxim group
Procedure: Rectal swab — Rectal swab every 3 days during hospitalization and then 30 days after the first antibiotic infusion
Drug: Cefotaxime/ceftriaxone — ceftriaxone or cefotaxime infusion at the discretion of the prescribing physician
  Arms: Cefotaxime or ceftriaxone group

SUMMARY:
The aim of this study was to compare the frequency of occurrence of digestive carrying of 3rd generation cephalosporin-resistant enterobacteriaceae (EB C3G-R), acquired during hospitalization in one of the participating departments, between patients treated with ceftriaxone and patients treated with cefotaxime

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Indication for antibiotic treatment with a 3rd generation injectable cephalosporin (cefotaxime or ceftriaxone)
* Signed Informed Consent

Exclusion Criteria:

* Hypersensitivity to ceftriaxone or cefotaxime, to another cephalosporin or to any of the excipients of the specialities concerned.
* History of severe hypersensitivity (e.g., anaphylactic reaction) to another class of antibacterial agent of the beta-lactam family (penicillins, monobactams and carbapenes)
* Subcutaneous administration of ceftriaxone
* Pregnant and breastfeeding woman
* Suspicion of Pseudomonas infection or documented Pseudomonas infection requiring ceftazidime treatment
* Suspicion of group III enterobacteriaceae infection or group III enterobacteriaceae infection requiring cefepime treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-04-03 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of occurrence of digestive carrying of EB C3G-R | 30 days after inclusion
  Frequency of occurrence of digestive carrying of EB C3G-R

SECONDARY OUTCOMES:
incidence rate of EB C3G-R infections | 2 years
  Evaluate the effect of systematic use of cefotaxime rather than ceftriaxone on the incidence rate of EB C3G-R infections in participating departments.
number of patients with occurrence of positive rectal swab with 3rd generation cephalosporin-resistant enterobacteriaceae (EB C3G-R) | 30 days after inclusion
  Compare the number of patients with occurrence of positive rectal swab with 3rd generation cephalosporin-resistant enterobacteriaceae (EB C3G-R), 30 days after inclusion, between patients treated with ceftriaxone and patients treated with cefotaxime.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France